CLINICAL TRIAL: NCT04739124
Title: Appropriation of the Connected Solution Freestyle Libre® in Adult Patients With Diabetes in the Context of Therapeutic Education
Acronym: APPRO-FSL
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PPRC11
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic patients: Patients presenting type 1 or type 2 diabetes, eligible for the prescription of Freestyle Libre
  Interventions: Other: Follow-up questionnaires; Other: Interviews
- Caregivers: Caregiver caring for diabetic patients and practicing therapeutic education on a regular basis
  Interventions: Other: Follow-up questionnaires

INTERVENTIONS:
Other: Follow-up questionnaires — The patient normally follows the education program as usual but research specific data is collected:
  * Biological sampling at the start and end of the education program (glycated hemoglobin).
  * Retrieval of usage and glycemic balance data from the Libreview online platform (at one week, one month and three months of use)
  * Iterative questionnaires allowing the study of factors of acceptance, appropriation and use (at the start of the study, at 4 weeks, at 12 weeks)
Other: Interviews — Semi-structured interviews will be carried out during the visits, either face-to-face or remotely.
  Groups: Diabetic patients

SUMMARY:
Following the proposal to self-monitor by the Freestyle Libre® (FSL) connected object, in diabetic patients in the context of therapeutic education, regarding the appropriation of FSL, what works, for which patients , in what specific contexts and by what mechanisms does it govern? A multicentric observational research will be conducted with mixed method design (follow-up using patient questionnaires) and semi-structured interviews of patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Patients

  * Have type 1 or type 2 diabetes (as included in the education program),
  * Be of legal age (over 18 years old),
  * Do not present legal protection measures due to incapacity (such as guardianship or guardianship).
  * Be able to read and speak French (elementary school level)
  * Be eligible for FSL prescription and authorize the sharing of your data in Libreview®
  * Be affiliated to a social security scheme
  * Have an email address or a phone allowing internet use
* Caregivers

  * Be registered on the roll of his professional order
  * Hold the certificate of 40 hours of training in therapeutic education.
  * Practice therapeutic education on a regular basis

Exclusion Criteria:

* Patients

  * presenting contraindications to the use of Freestyle Libre® (known allergies to adhesive products, coagulation disorders, not treated with insulin therapy or with less than 3 insulin injections per day or continuously, not requiring glycemic monitoring or less than 3 times a day)
  * Patient refusing to follow the education program,
  * Minors, patients under administrative or judicial supervision)
  * Pregnant women,
  * Patients who cannot be contacted in an emergency,
  * Persons in a position to give their consent but with an inability to read / write the French language.
  * Patients who do not have an email address or a phone allowing internet use.
* Caregivers

  * Failure to register with the professional order (except those of the Army Health Service who are exempt)
  * Non-possession of the 40-hour therapeutic education training certificate.
  * Not practicing FSL education

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of diabetic patients and their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Correlation between appropriation factors, intention to use, Freestyle Libre use and glycemic control | 3 months
  longitudinal multifactor analysis by structural equation modeling of the research model created specifically

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Avicenne, Bobigny
  - Hopital d'Instruction des Armées Bégin, Saint-Mandé

IPD SHARING:
Plan to Share IPD: Undecided